CLINICAL TRIAL: NCT00319904
Title: The Partners Genetics Collaborative Study of Schizophrenia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Daphne Holt, Associate Professor of Psychiatry, Massachusetts General Hospital
Other Study IDs: 2001-P-000560
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; DNA
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA is extracted and stored for future anaysis of genes that may be associated with schizophrenia
Oversight: Data Monitoring Committee: No

SUMMARY:
We will collect DNA from 500 rigorously diagnosed patients with schizophrenia to allow us in the future to examine phenotypic subtypes in relation to genetic variants. Phenotypes will include subgroups based on clinical symptoms, medication response, or other biological markers including neuroimaging or pharmacologic challenges.

DETAILED DESCRIPTION:
Specific Aims:

We will collect DNA from 500 rigorously diagnosed patients with schizophrenia to allow us in the future to examine phenotypic subtypes in relation to genetic variants. Phenotypes will include subgroups based on clinical symptoms, medication response, or other biological markers including neuroimaging or pharmacologic challenges.

Subjects:

DNA samples and clinical characterization will be obtained from 500 schizophrenia patients treated at the Freedom Trail Clinic of the Erich Lindemann Mental Health Association and the MGH First Episode Psychosis Program.

The diagnostic interview will be conducted by a research psychiatrist and will typically take between 1-3 hours. The following clinical data will be obtained for all subjects:

Demographics (age, gender, ethnicity) Weight, height Current medications and doses Age of onset (prodrome and psychosis) Incidence of psychotic disorders in first-degree family members (without identifiers) Diagnosis with subtype History of hallucinations, delusions, negative symptoms, disorganization and mood disorder History of response (full, partial, or no response) of symptoms (hallucinations, delusions, disorganization and negative symptoms) to conventional antipsychotics, atypicals or clozapine Number of hospitalizations Smoking behaviors (using the Fagerstrom)

The additional clinical assessment will take approximately 2-3 hours and will include the following clinical rating scales and cognitive tests:

Symptom Rating Scales:

Positive and Negative Symptom Scale (PANSS) Scale for Assessment of Negative Symptoms (SANS) Abnormal Involuntary Movements Scale (AIMS) (examination) Clinical Global Impressions-Severity of Illness Scale (CGI) (observational) Beck Depression Inventory (BDI-II) Simpson-Angus Scale (SAS)

Cognitive Battery:

Wechsler Adult Intelligence Scale (selected subtests) (WAIS-III) North American Adult Reading Test (NAART) Stroop Test Wisconsin Card Sorting Test (WCST) California Verbal Learning Test (CVLT) Verbal Fluency (FAS) Finger Tapping CPT-IP

Collection of Blood Samples:

Four tubes of blood will be drawn from an antecubital vein from each participant using an EDTA and non-EDTA vacutainers. Tubes will be labeled with the study, date, and an encrypted identification of the subject. Samples will be used for DNA extraction and measurement of serum and RBC folate and homocysteine.

Genetic Analysis:

Genes will be studied that have been identified in linkage studies of patients with schizophrenia that have compelling biology relevant to potential mechanisms of etiology or drug response. Approximately 20 candidate genes have been identified with varying levels of evidence-this number is rapidly expanding. We will review the potential list of candidate genes when we have completed collecting the sample and will identify the most promising genotypic targets for analysis. If approved by the IRB, comparisons with other populations (such as depressed patients or nonpsychiatric controls) may be performed in collaboration with other investigators.

Risks:

While the clinical assessment may be stressful, the questions contained in the diagnostic instruments do not differ from those asked in routine clinical evaluations. Phlebotomy may produce discomfort, bruising, and rarely, infection. In theory, release of genetic information to patients could be upsetting and release to other parties could represent a serious breach of privacy. Extensive precautions will be taken to prevent such an occurrence.

All DNA analyses will be performed on anonymous samples.

Subject Remuneration:

Subjects who agree to phlebotomy and complete the psychiatric evaluation will be remunerated $25 for their time. Subjects who complete the additional cognitive battery and clinical rating scales will be remunerated a total of $50 for their time.

ELIGIBILITY:
Inclusion Criteria:

Schizophrenia, any subtype Ages 18-70 years Males or females English speaking Ability to complete symptom rating scales and cognitive tests Ability to provide informed consent

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2001-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
phenotypic subtypes in relation to genetic variants | Baseline
  We will collect DNA from 500 patients with schizophrenia to examine phenotypic subtypes in relation to genetic variants. Phenotypes will include subgroups based on clinical symptoms, medication response, or other biological markers including neuroimaging or pharmacologic challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne J Holt, M.D., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Result] Roffman JL, Gollub RL, Calhoun VD, Wassink TH, Weiss AP, Ho BC, White T, Clark VP, Fries J, Andreasen NC, Goff DC, Manoach DS. MTHFR 677C --> T genotype disrupts prefrontal function in schizophrenia through an interaction with COMT 158Val --> Met. Proc Natl Acad Sci U S A. 2008 Nov 11;105(45):17573-8. doi: 10.1073/pnas.0803727105. Epub 2008 Nov 6. PMID 18988738